CLINICAL TRIAL: NCT04719221
Title: A Single-center, Randomized, Parallel-group, Open-label Pilot Study to Evaluate the Impact of Evolocumab as an Additional Lipid-lowering Therapy to Changes in Lipid Core Burden Index of Non-culprit Vulnerable Plaque in Patients Who Underwent Percutaneous Coronary Intervention for the Acute Coronary Syndrome
Brief Title: Impact of Evolocumab as an Additional Lipid-lowering Therapy to Changes in Lipid Core Burden Index of Non-culprit Vulnerable Plaque in Patients Who Underwent Percutaneous Coronary Intervention for the Acute Coronary Syndrome
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Korea University Anam Hospital (Other)
Responsible Party: Principal Investigator, Jung-Joon Cha, Assistant Professor, Korea University Anam Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ELoNirs-ACS
Record Dates: First submitted 2021-01-12; First posted 2021-01-22 (Actual); Last update posted 2023-10-05 (Actual); Status verified 2023-10

CONDITIONS: Clinical Trial; Acute Coronary Syndrome
Keywords: evolocumab; Spectroscopy, Near-Infrared
MeSH Terms: conditions — Acute Coronary Syndrome | interventions — evolocumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Statin+Ezetimibe (Placebo Comparator): Drug: Statin + Ezetimibe (combined cholesterol therapy)
  Interventions: Drug: Evolocumab; Device: NIRS IVUS
- Statin+Ezetimibe+Evolocumab (Active Comparator): Drug: Statin + Ezetimibe (combined cholesterol therapy) and Drug: Evolocumab
  Interventions: Drug: Evolocumab; Device: NIRS IVUS

INTERVENTIONS:
Drug: Evolocumab — The maximum dose of combined cholesterol therapy (Statin + Ezetimibe) is prescribed for 2 months, and a cholesterol test is performed in an outpatient clinic to ensure that LDL-Cholesterol <70mg/dL is met. Patients who do not meet the criteria are randomized to maintain current treatment or receive additional Evolocumab according to randomization.
  Other Names: Repatha
Device: NIRS IVUS — near-infrared spectroscopy

SUMMARY:
This study aimed to investigate the impact of intensive cholesterol-lowering therapy (including evolocumab), drug treatment for high-risk plaques (Vulnerable plaques) with a high probability of developing acute coronary syndrome. The purpose of this study is to determine the effect of the change in the Lipid core burden index and compare the rate of cardiac events over 12 months following cholesterol therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Over 19 years old
2. Patients who agree to the study plan and clinical follow-up plan, voluntarily decide to participate in this study, and consent in writing to the consent to use information
3. Patients who underwent NIRS-IVUS guided coronary stent surgery for acute coronary syndrome
4. Patients who did not meet the LDL-Cholesterol level (<70mg/dL) even after receiving the maximum dose of combined cholesterol therapy for 2 months

Exclusion Criteria:

1. Subjects with known hypersensitivity or contraindications to the following drugs or substances: heparin, aspirin, clopidogrel, ticagrelor, prasugrel, rosuvastatin, ezetimibe, evolocumab, lansoprazole, cobalt chromium, stainless steel nickel And contrast agents (however, even a subject who is hypersensitive to contrast agents can register if they can be controlled by steroids and pheniramine, except for known anaphylaxis.)
2. Pregnant women, lactating women, or women of childbearing age who plan to become pregnant during this study
3. Subjects who plan to have surgery to stop antiplatelet drugs within 12 months from registration
4. Those whose surviving life is expected to be less than 1 year
5. Subjects who visited the hospital due to psychogenic shock and are predicted to have low survival probability based on medical judgment
6. Subjects participating in a randomized study on cholesterol therapy

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-03-01 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Change of 1-year lipid core burden index | 1 year

SECONDARY OUTCOMES:
patient-oriented composite end point | 1 year
  composite of all cause mortality, any myocardial infarction, and any revascularization
Percentage of All cause mortality | 1 year
Percentage of cardiac death | 1 year
Percentage of myocardial infarction | 1 year
Percentage of revascularization | 1 year
Rate of usage of cholesterol lowering agents (2 month) | 1 year
Rate of usage of cholesterol lowering agents (12 month) | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Korea University Anam Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Levine GN, Bates ER, Blankenship JC, Bailey SR, Bittl JA, Cercek B, Chambers CE, Ellis SG, Guyton RA, Hollenberg SM, Khot UN, Lange RA, Mauri L, Mehran R, Moussa ID, Mukherjee D, Nallamothu BK, Ting HH; American College of Cardiology Foundation; American Heart Association Task Force on Practice Guidelines; Society for Cardiovascular Angiography and Interventions. 2011 ACCF/AHA/SCAI Guideline for Percutaneous Coronary Intervention. A report of the American College of Cardiology Foundation/American Heart Association Task Force on Practice Guidelines and the Society for Cardiovascular Angiography and Interventions. J Am Coll Cardiol. 2011 Dec 6;58(24):e44-122. doi: 10.1016/j.jacc.2011.08.007. Epub 2011 Nov 7. No abstract available. PMID 22070834
- [Background] Bashore TM, Balter S, Barac A, Byrne JG, Cavendish JJ, Chambers CE, Hermiller JB Jr, Kinlay S, Landzberg JS, Laskey WK, McKay CR, Miller JM, Moliterno DJ, Moore JW, Oliver-McNeil SM, Popma JJ, Tommaso CL; ACCF Task Force Members. 2012 American College of Cardiology Foundation/Society for Cardiovascular Angiography and Interventions expert consensus document on cardiac catheterization laboratory standards update: A report of the American College of Cardiology Foundation Task Force on Expert Consensus documents developed in collaboration with the Society of Thoracic Surgeons and Society for Vascular Medicine. J Am Coll Cardiol. 2012 Jun 12;59(24):2221-305. doi: 10.1016/j.jacc.2012.02.010. Epub 2012 May 8. No abstract available. PMID 22575325
- [Background] Moussa I, Hermann A, Messenger JC, Dehmer GJ, Weaver WD, Rumsfeld JS, Masoudi FA. The NCDR CathPCI Registry: a US national perspective on care and outcomes for percutaneous coronary intervention. Heart. 2013 Mar;99(5):297-303. doi: 10.1136/heartjnl-2012-303379. Epub 2013 Jan 15. PMID 23322530
- [Background] Task Force Members; Montalescot G, Sechtem U, Achenbach S, Andreotti F, Arden C, Budaj A, Bugiardini R, Crea F, Cuisset T, Di Mario C, Ferreira JR, Gersh BJ, Gitt AK, Hulot JS, Marx N, Opie LH, Pfisterer M, Prescott E, Ruschitzka F, Sabate M, Senior R, Taggart DP, van der Wall EE, Vrints CJ; ESC Committee for Practice Guidelines; Zamorano JL, Achenbach S, Baumgartner H, Bax JJ, Bueno H, Dean V, Deaton C, Erol C, Fagard R, Ferrari R, Hasdai D, Hoes AW, Kirchhof P, Knuuti J, Kolh P, Lancellotti P, Linhart A, Nihoyannopoulos P, Piepoli MF, Ponikowski P, Sirnes PA, Tamargo JL, Tendera M, Torbicki A, Wijns W, Windecker S; Document Reviewers; Knuuti J, Valgimigli M, Bueno H, Claeys MJ, Donner-Banzhoff N, Erol C, Frank H, Funck-Brentano C, Gaemperli O, Gonzalez-Juanatey JR, Hamilos M, Hasdai D, Husted S, James SK, Kervinen K, Kolh P, Kristensen SD, Lancellotti P, Maggioni AP, Piepoli MF, Pries AR, Romeo F, Ryden L, Simoons ML, Sirnes PA, Steg PG, Timmis A, Wijns W, Windecker S, Yildirir A, Zamorano JL. 2013 ESC guidelines on the management of stable coronary artery disease: the Task Force on the management of stable coronary artery disease of the European Society of Cardiology. Eur Heart J. 2013 Oct;34(38):2949-3003. doi: 10.1093/eurheartj/eht296. Epub 2013 Aug 30. No abstract available. PMID 23996286
- [Background] Nallamothu BK, Tommaso CL, Anderson HV, Anderson JL, Cleveland JC Jr, Dudley RA, Duffy PL, Faxon DP, Gurm HS, Hamilton LA, Jensen NC, Josephson RA, Malenka DJ, Maniu CV, McCabe KW, Mortimer JD, Patel MR, Persell SD, Rumsfeld JS, Shunk KA, Smith SC Jr, Stanko SJ, Watts B. ACC/AHA/SCAI/AMA-Convened PCPI/NCQA 2013 Performance Measures for Adults Undergoing Percutaneous Coronary Intervention: A Report of the American College of Cardiology/American Heart Association Task Force on Performance Measures, the Society for Cardiovascular Angiography and Interventions, the American Medical Association-Convened Physician Consortium for Performance Improvement, and the National Committee for Quality Assurance. Circulation. 2014 Feb 25;129(8):926-49. doi: 10.1161/01.cir.0000441966.31451.3f. Epub 2013 Dec 19. No abstract available. PMID 24357402
- [Background] Authors/Task Force members; Windecker S, Kolh P, Alfonso F, Collet JP, Cremer J, Falk V, Filippatos G, Hamm C, Head SJ, Juni P, Kappetein AP, Kastrati A, Knuuti J, Landmesser U, Laufer G, Neumann FJ, Richter DJ, Schauerte P, Sousa Uva M, Stefanini GG, Taggart DP, Torracca L, Valgimigli M, Wijns W, Witkowski A. 2014 ESC/EACTS Guidelines on myocardial revascularization: The Task Force on Myocardial Revascularization of the European Society of Cardiology (ESC) and the European Association for Cardio-Thoracic Surgery (EACTS)Developed with the special contribution of the European Association of Percutaneous Cardiovascular Interventions (EAPCI). Eur Heart J. 2014 Oct 1;35(37):2541-619. doi: 10.1093/eurheartj/ehu278. Epub 2014 Aug 29. No abstract available. PMID 25173339
- [Background] Madder RD, Goldstein JA, Madden SP, Puri R, Wolski K, Hendricks M, Sum ST, Kini A, Sharma S, Rizik D, Brilakis ES, Shunk KA, Petersen J, Weisz G, Virmani R, Nicholls SJ, Maehara A, Mintz GS, Stone GW, Muller JE. Detection by near-infrared spectroscopy of large lipid core plaques at culprit sites in patients with acute ST-segment elevation myocardial infarction. JACC Cardiovasc Interv. 2013 Aug;6(8):838-46. doi: 10.1016/j.jcin.2013.04.012. Epub 2013 Jul 17. PMID 23871513
- [Background] Madder RD, Steinberg DH, Anderson RD. Multimodality direct coronary imaging with combined near-infrared spectroscopy and intravascular ultrasound: initial US experience. Catheter Cardiovasc Interv. 2013 Feb;81(3):551-7. doi: 10.1002/ccd.23358. Epub 2012 Jan 10. PMID 22110009
- [Background] Puri R, Madder RD, Madden SP, Sum ST, Wolski K, Muller JE, Andrews J, King KL, Kataoka Y, Uno K, Kapadia SR, Tuzcu EM, Nissen SE, Virmani R, Maehara A, Mintz GS, Nicholls SJ. Near-Infrared Spectroscopy Enhances Intravascular Ultrasound Assessment of Vulnerable Coronary Plaque: A Combined Pathological and In Vivo Study. Arterioscler Thromb Vasc Biol. 2015 Nov;35(11):2423-31. doi: 10.1161/ATVBAHA.115.306118. Epub 2015 Sep 3. PMID 26338299
- [Background] Stone GW, Maehara A, Muller JE, Rizik DG, Shunk KA, Ben-Yehuda O, Genereux P, Dressler O, Parvataneni R, Madden S, Shah P, Brilakis ES, Kini AS; CANARY Investigators. Plaque Characterization to Inform the Prediction and Prevention of Periprocedural Myocardial Infarction During Percutaneous Coronary Intervention: The CANARY Trial (Coronary Assessment by Near-infrared of Atherosclerotic Rupture-prone Yellow). JACC Cardiovasc Interv. 2015 Jun;8(7):927-36. doi: 10.1016/j.jcin.2015.01.032. Epub 2015 May 20. PMID 26003018
- [Background] Kini AS, Vengrenyuk Y, Shameer K, Maehara A, Purushothaman M, Yoshimura T, Matsumura M, Aquino M, Haider N, Johnson KW, Readhead B, Kidd BA, Feig JE, Krishnan P, Sweeny J, Milind M, Moreno P, Mehran R, Kovacic JC, Baber U, Dudley JT, Narula J, Sharma S. Intracoronary Imaging, Cholesterol Efflux, and Transcriptomes After Intensive Statin Treatment: The YELLOW II Study. J Am Coll Cardiol. 2017 Feb 14;69(6):628-640. doi: 10.1016/j.jacc.2016.10.029. Epub 2016 Oct 29. PMID 27989886
- [Background] Kini AS, Baber U, Kovacic JC, Limaye A, Ali ZA, Sweeny J, Maehara A, Mehran R, Dangas G, Mintz GS, Fuster V, Narula J, Sharma SK, Moreno PR. Changes in plaque lipid content after short-term intensive versus standard statin therapy: the YELLOW trial (reduction in yellow plaque by aggressive lipid-lowering therapy). J Am Coll Cardiol. 2013 Jul 2;62(1):21-9. doi: 10.1016/j.jacc.2013.03.058. Epub 2013 May 1. PMID 23644090
- [Background] Stone GW, Maehara A, Ali ZA, Held C, Matsumura M, Kjoller-Hansen L, Botker HE, Maeng M, Engstrom T, Wiseth R, Persson J, Trovik T, Jensen U, James SK, Mintz GS, Dressler O, Crowley A, Ben-Yehuda O, Erlinge D; PROSPECT ABSORB Investigators. Percutaneous Coronary Intervention for Vulnerable Coronary Atherosclerotic Plaque. J Am Coll Cardiol. 2020 Nov 17;76(20):2289-2301. doi: 10.1016/j.jacc.2020.09.547. Epub 2020 Oct 15. PMID 33069847
- [Background] Pu J, Mintz GS, Brilakis ES, Banerjee S, Abdel-Karim AR, Maini B, Biro S, Lee JB, Stone GW, Weisz G, Maehara A. In vivo characterization of coronary plaques: novel findings from comparing greyscale and virtual histology intravascular ultrasound and near-infrared spectroscopy. Eur Heart J. 2012 Feb;33(3):372-83. doi: 10.1093/eurheartj/ehr387. Epub 2011 Oct 20. PMID 22019821